CLINICAL TRIAL: NCT06142435
Title: Mild Traumatic Brain Injury Identification and Monitoring Through Retional Scanning
Brief Title: mTBI Identification and Monitoring Through Retinal Scanning
Status: Recruiting | Type: Observational
Sponsor: Rebiscan, Inc. (Industry)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: BU-001
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be drawn by venipuncture, collected in Serum Separator Tubes, clotted for 30-60 min, centrifuged at 1,500 rpm for 15 min, and stored at -80°C until batch analysis for serum levels of four well-established brain injury biomarkers (i.e., astrocyte-derived glial fibrillary acidic protein; GFAP; neuron-derived ubiquitin carboxy-terminal hydrolyzing enzyme L1, UCH-L1; neuron-derived total microtubule-associated protein tau, T-Tau; neuron-derived neurofilament-light chain, NF-L) using the Quanterix SIMOA Neurology 4-plex "B" kit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Controls: Participants should not be part of the Intended Use Population. Subjects that present to the hospital, clinic, or emergency department, either as a patient or non-patient, with no history of head trauma and, are 18-45 years of age.
  Interventions: Device: Head and Intraocular Trauma Tool
- TBI-Suspected Patients: TBI participants 18-45 years of age, recruited from patients at a clinical research facility who present with head trauma. Clinical evaluation for the patient can be positive (target condition present) or negative (target condition absent) for mTBI. Testing will occur on Day-0, Day-14, and Day-30.
  Interventions: Device: Head and Intraocular Trauma Tool

INTERVENTIONS:
Device: Head and Intraocular Trauma Tool — HITT device to scan the eyes of participants up to 3 times (~45 seconds each) at the time of admittance to study. The participant is to place the chin in the chin-rest and fixate on the illuminated light on the device.
  Other Names: HITT

SUMMARY:
Rebion has developed a device, the Rebion trauma tool (referred to as the head and intraocular trauma tool, or "HITT"), that detects ocular fixation and alignment using a binocular retinal scan. Preliminary data obtained from hospitalized patients with a clinically-confirmed traumatic brain injury (TBI) and uninjured controls indicates that the device can detect changes in ocular fixation, alignment, and saccades that are related to brain injury. This study seeks to evaluate the ability of the Rebion trauma tool to assess perturbations in eye movements resulting from TBI. The study will enroll 60 TBI patients and 20 controls.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years
2. Presents to the facility within 2 weeks of head trauma
3. Able to provide informed consent

   * If minor, then able to provide parental consent and minor consent
4. Able to participate in the examination, including the ability to follow simple instructions
5. Fluency in English or Spanish

Exclusion Criteria:

1. Glasgow Coma Scale score equal to or less than 13 at the time of study enrollment
2. Under the influence of alcohol or drugs
3. Previous eye surgery
4. Visual acuity known to be 20/200 or less in either eye
5. Known strabismus, amblyopia (lazy eye), or double vision
6. Known eye movement disorder, including nystagmus
7. Known optic nerve disease, including papilledema or optic neuropathy
8. Known retinal disease, including macular degeneration or retinal degeneration
9. Known cataract
10. History of neurosurgery
11. History of stroke/brain hemorrhage, brain tumor, or epilepsy
12. Any head trauma requiring medical attention from a physician within the last 6 months
13. Diagnosed dementia or cognitive impairment requiring assistance for daily living
14. Other condition(s) under the care of a neurologist
15. Psychiatric hospitalization in the last 90 days
16. Subject considered unsuitable for participation in this clinical trial by PI, treating clinician, or study research staff
17. Any minor brain injury regardless of loss of consciousness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population includes target participants that enroll within two weeks of blunt head trauma, with a Glasgow Coma Scale score equal to or greater than thirteen, A minimum of sixty Target Condition subjects will be enrolled. All studies will be complete within thirty days of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
TBI Detection | 1 day
  Patients who present with suspected TBI to the clinic will have their eyes scanned to identify whether the HITT device can accurately identify patients with TBI.

SECONDARY OUTCOMES:
TBI Monitor | 14 days
  Patients who present with suspected TBI to the clinic and had initially been tested for TBI detection will receive a second set of scans at 2 weeks to identify whether the HITT device can accurately identify patients with TBI.
TBI Monitor | 30 days
  Patients who present with suspected TBI to the clinic and had initially been tested for TBI detection will receive a second set fo scans at one month to identify whether the HITT device can accurately identify patients with TBI.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Medical Center Concussion Clinic, Ryan Center for Sports Medicine & Rehabilitation at Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate data and individual test reports will be made available to the HITT device manufacturer to better understand its performance at identifying TBI. Personally-identifiable data will not be shared with anyone outside of the Boston Medical Center.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be shared on an ongoing basis, and cumulatively at the end of the study. Study length is expected to be 2 months from the first enrolled participant.
Access Criteria: Data will only be shared with researchers involved in the study at the Boston Medical Center, and only trained staff members at the device manufacturer.